CLINICAL TRIAL: NCT00329316
Title: Prevention of Recurrent Preterm Delivery by a Natural Progesterone Agent
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn for financial problems. We didnwt get a grant we needed for purchesing the medication for the study.
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: PTL Progesterone Perlitz.CTIL
Record Dates: First submitted 2006-05-23; First posted 2006-05-24 (Estimated); Last update posted 2008-06-27 (Estimated); Status verified 2007-06

CONDITIONS: Pregnancy; Premature Birth
Keywords: Pre-term labor; progesterone
MeSH Terms: conditions — Premature Birth

INTERVENTIONS:
Drug: Crinone Gel 8%

SUMMARY:
To examine the preterm delivery rate of a preterm delivery high risk group of pregnant women, using once daily natural progesterone agent.

ELIGIBILITY:
Inclusion Criteria:

Pregnancy 24 weeks' gestation Preterm labor in previous pregnancies

-

Exclusion Criteria:

* No medications for PTL or any kind of progesterone.
* Cervical suture
* Multiple pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Yuri Perlitz, MD, Study Chair — The Baruch Padeh Medical Center, Poriya; Mosheh Ben Ami, Prof., Principal Investigator — Head of Obs/Gyn ,The Baruch Padeh Medical center, Poriya